**Nombre del estudio:** El efecto de participar en charlas de planificación sobre la atención médica anticipada (ENACT, siglas en inglés). Visitas grupales de intervención en la atención primaria para los adultos mayores con y sin enfermedad de Alzheimer

Investigadora Principal: Hillary D. Lum, MD, PhD

Núm. de COMIRB: 20-1978 Versión fechada: 7.10.2023

### ¿De qué se trata este estudio?

Este estudio pretende obtener más información acerca de cómo mejorar la planificación anticipada de la atención médica para los pacientes a través de su clínica de atención primaria.

Se le pide participar en este estudio ÚNICAMENTE porque usted o su ser querido reciben atención primaria aquí. Usted <u>NO</u> fue elegido para participar en este estudio debido a algún problema médico que pudieran tener usted o su ser querido. Tampoco fue elegido porque su médico o los médicos que dirigen este estudio creen que necesita usted llenar estos formularios.

## ¿Qué le pide hacer este estudio?

## Si decide participar en este estudio, y como paciente:

- 1. Se le preguntará acerca de su experiencia con la planificación anticipada del cuidado médico y se le pedirá su punto de vista acerca de su salud. Se estima que las encuestas tomarán entre 20-30 minutos. Le haremos preguntas breves para evaluar su memoria. El personal del estudio le informará su puntaje en la valoración de memoria y lo que se considera un puntaje normal. Los resultados del examen de memoria no se utilizan para hacer un diagnóstico.
- 2. Después de las encuestas, se le seleccionará sin seguir ningún orden en particular (al azar), para recibir información sobre la planificación anticipada de la atención médica, de una de las siguientes maneras:
  - a) Recibirá por correo postal, información de la planificación anticipada de la atención médica.
  - b) Recibirá por correo postal, información de la planificación anticipada de la atención médica y dos visitas médicas grupales, con un mes de diferencia entre cada visita. Las visitas se harán en la clínica de atención primaria. Aproximadamente participará con 8-10 pacientes que también forman parte del estudio. Cada visita grupal durará alrededor de 2 horas. Cada visita grupal ofrece apoyo, educación, y

conversación sobre la planificación anticipada del cuidado médico. Las visitas grupales serán grabadas en video-audio. Esto nos permite estudiar cómo funciona la intervención de las visitas grupales. Las grabaciones no se distribuirán ni se utilizarán para ningún otro propósito que no sea el estudio de investigación.

Si usted es seleccionado para recibir información acerca de la planificación del cuidado médico anticipado, en la opción que incluye las visitas médicas grupales, deberá dar su copago regular que aplica bajo su seguro médico, ya que las visitas se consideran parte de su cuidado médico.

- 3. Seis meses después de unirse al estudio, nos comunicaremos con usted por teléfono para hacerle algunas preguntas breves acerca de su experiencia. La llamada tomará entre 20-30 minutos.
- 4. También a los seis meses, invitaremos a algunos participantes a tomar parte en una entrevista voluntaria ya sea por teléfono o video, para saber qué funcionó y qué no funcionó en la visita grupal. Las entrevistas podrían durar entre 20-30 minutos.
- 5. El personal del estudio tomará datos de su expediente médico para utilizarlos en el estudio. La información que lo puede identificar (por ej. su nombre, dirección, y fecha de nacimiento) no se incluirá en las publicaciones.

En seis meses, después de que se haya terminado el estudio y haya usted recibido por correo la información acerca de la planificación del cuidado médico anticipado, usted podrá elegir participar en las visitas médicas grupales que tienen que ver con la planificación anticipada del cuidado médico, como parte de su atención médica regular.

# Si usted se une a este estudio, y es una <u>persona que brinda apoyo o</u> que cuida al paciente:

1. Le pediremos que conteste las preguntas de unas encuestas cortas relacionadas con su parentesco con el paciente, y a preguntas sobre su información demográfica. Hemos calculado que las encuestas tomarán unos 5 minutos.

- 2. Se le invitará a participar en el estudio junto al paciente, quien será seleccionado al azar para recibir información sobre la planificación del cuidado médico anticipado, de una de las siguientes maneras:
  - a) Recibirá por correo información sobre la planificación anticipada del cuidado médico
  - b) Recibirá por correo información sobre la planificación anticipada del cuidado médico, y también asistirá a dos visitas médicas grupales en la clínica de atención primaria del paciente, participando como persona de apoyo u observador. Este grupo no forma parte de su cuidado clínico. Las visitas en grupo serán grabadas en video-audio.
- 3. Seis meses después de unirse al estudio, se invitará a algunas personas a participar en una entrevista voluntaria por teléfono o video para saber qué funcionó y qué no funcionó en la visita grupal. Las entrevistas podrían durar entre 20-30 minutos.

### Cuáles son los posibles riesgos o efectos secundarios:

- 1. Incomodidad psicológica: Algunas personas pueden sentirse incómodas al pensar o hablar sobre la planificación anticipada del cuidado médico o sobre los problemas relacionados con los últimos días de vida. Si llegara usted a sentirse incómodo, puede dejar de revisar el material sobre el tema, o dejar de participar en las visitas grupales y dejar de responder a las preguntas en cuanto lo desee. Algunos pacientes también podrían sentir incomodidad durante la evaluación de la memoria.
- 2. Pérdida de confidencialidad: En todos los estudios se corre el riesgo de perder cierta privacidad. Haremos todo lo posible por proteger su privacidad y confidencialidad. Si forma parte de la visita grupal, les recordaremos a todos los participantes la importancia de mantener la privacidad de los demás participantes. Los registros de su estudio se mantendrán seguros en unidades informáticas electrónicas seguras y se destruirán al final del estudio.
- 3. Podría haber otros riesgos no evidentes para los investigadores.

La participación en este estudio es voluntaria. Usted tiene la opción de formar parte del estudio. No tiene que participar si no lo desea. También puede decidir, en cualquier momento, dejar de ser un participante activo. Si así lo decide, dejaremos de contactarlo. Continuaremos recopilando información de su expediente médico para utilizarla en el estudio, excepto

si usted informa por escrito a la Dra. Hillary Lum a la siguiente dirección o correo electrónico:

Hillary Lum, MD, PhD 12631 East 17<sup>th</sup> Ave Mail Stop B-179 Aurora, CO 80045 Hillary.Lum@cuanschutz.edu

Si es un paciente, se le ofrecerá una tarjeta de regalo de \$25 por completar la primera parte del studio y otra tarjeta de regalo de \$25 por completar la encuesta de 6 meses.

Si es usted un cuidador y se le solicita participar en una entrevista, se le ofrecerá una tarjeta de regalo de \$25.

Si usted u otra persona comparten información sobre algún incidente que haya sucedido, el cual estamos legalmente obligados a reportar, lo reportaremos (por ej., abuso a personas de la tercera edad).

Este estudio no está diseñado para beneficiarlo directamente. Esta investigación está siendo financiada por el Instituto Nacional del Envejecimiento.

## Privacidad y confidencialidad

La información que colectemos será utilizada para este estudio, y a la vez, puede ser importante para investigaciones futuras. Su información podría utilizarse para investigaciones futuras o distribuirse a otros investigadores para estudios futuros, sin un consentimiento adicional, si se elimina la información que lo identifica.

Mantendremos confidencial su participación en este estudio de investigación en la medida permitida por la ley. Sin embargo, es posible que otras personas se den cuenta de su participación en este estudio. Por ejemplo, las siguientes personas/grupos pueden inspeccionar y copiar registros relacionados con esta investigación.

- La Oficina de Protección de Investigaciones Humanas en el Departamento de Salud y Servicios Humanos de los Estados Unidos
- La Junta de Revisión Institucional Múltiple de Colorado (un comité que revisa y aprueba los estudios de investigación)
- El patrocinador del estudio, los Institutos Nacionales de la Salud

Algunos de estos registros pueden contener información que lo identifica personalmente. Haremos todo esfuerzo razonable por mantener, privada y confidencial, la información personal en su registro de investigación, pero no le podemos garantizar la confidencialidad absoluta.

Este estudio ha recibido un Certificado de Confidencialidad de parte del gobierno federal el cual ayuda a proteger su privacidad. El Certificado les prohíbe a los investigadores revelar su nombre, y cualquier información o documento de la investigación que lo identifique. Un certificado de este tipo, protege de ser revelada, la información del estudio en procesos civiles a nivel federal, estatal o local, al igual que en otros procesos criminales, administrativos o legislativos. Las protecciones aplican solamente a sus registros del estudio de investigación.

**Si tiene alguna pregunta**, comuníquese en todo momento con la Dra. Hillary Lum al (303) 724-1911. Asimismo, si tiene preguntas acerca de sus derechos como participante en el estudio, llame al COMIRB (el Consejo de Revisión Institucional responsable) al (303) 724-1055.

Nos gustaría contactarlo para inscribirlo en investigaciones futuras: Si está de acuerdo, nos gustaría utilizar la información que recopilamos en este estudio para determinar si es elegible para estudios futuros de investigación. Si acepta, agregaremos su nombre a una base de datos que se utilizará para enlistar a participantes para estudios de investigación. Si no acepta, no lo agregaremos a la base de datos mencionada, ni tampoco nos pondremos en contacto con usted sobre otras oportunidades de estudios de investigación.

Por último, puede usted revocar su autorización para ser contactado para estudios futuros en cualquier momento que lo desee. Si desea hacerlo, llame a la Dra. Hillary Lum al (303) 724-1911 e infórmele que ya no desea ser contactado para estudios de investigación.